CLINICAL TRIAL: NCT04374877
Title: A Phase 1/1b Study of CHS-388 (Formerly Known as SRF388) in Patients With Advanced Solid Tumors
Brief Title: Study of CHS-388 (Formerly Known as SRF388) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRF388-101; KEYNOTE-C16 (Other: Merck Sharp & Dohme LLC); MK-3475-C16 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Clear Cell Renal Cell Carcinoma; Hepatocellular Carcinoma; Non-small Cell Lung Cancer
Keywords: metastatic solid tumors; advanced solid tumors; Phase 1; CHS-388; IL-27; safety; efficacy; immunotherapy; cancer; immuno-oncology; kidney cancer; renal cell carcinoma; liver cancer; hepatocellular carcinoma; non-small cell lung cancer; pembrolizumab; PD-1; toripalimab; SRF388
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Neoplasms; Kidney Neoplasms; Liver Neoplasms | interventions — pembrolizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A Monotherapy Dose Escalation (Experimental): The Part A monotherapy dose escalation portion of the study will evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of CHS-388 as monotherapy in up to 30 patients with advanced solid tumors.
  Interventions: Drug: CHS-388
- Part B CHS-388 Monotherapy Expansion (Experimental): Part B monotherapy expansion will evaluate the safety, tolerability, PK, pharmacodynamics, and efficacy of CHS-388 monotherapy at the recommended phase 2 dose (RP2D) in up to 40 patients with ccRCC, up to 40 patients with HCC, and up to 40 patients with NSCLC.
  Interventions: Drug: CHS-388
- Part C CHS-388 in Combination with Pembrolizumab (Experimental): Part C will evaluate the safety, preliminary efficacy, tolerability, and PK of CHS-388 in combination with pembrolizumab in patients with advanced RCC or HCC, or anti-PD(L)1 relapsed/refractory advanced NSCLC.
  Interventions: Drug: CHS-388; Drug: Pembrolizumab
- Part D CHS-388 in Combination with Toripalimab (Experimental): Part D will evaluate the safety, preliminary efficacy, tolerability, and PK of CHS-388 in combination with toripalimab in patients with anti-PD(L)1 relapsed/refractory advanced NSCLC.
  Interventions: Drug: CHS-388; Drug: Toripalimab

INTERVENTIONS:
Drug: CHS-388 — CHS-388 is a fully human IgG1 antibody against IL-27. Inhibition of IL-27 with CHS-388 reduces STAT1 phosphorylation leading to increased pro-inflammatory (anti-tumor) cytokine secretion (e.g., IFN-g, TNF-a) and decreased expression of inhibitory immune checkpoint receptors (e.g., PD-L1, TIGIT, LAG3) on immune cells that may result in anticancer therapeutic activity.
  Other Names: Casdozokitug
Drug: Pembrolizumab — Pembrolizumab by intravenous (IV) infusion
  Other Names: Keytruda®
  Arms: Part C CHS-388 in Combination with Pembrolizumab
Drug: Toripalimab — Toripalimab by IV infusion
  Other Names: Loqtorzi®
  Arms: Part D CHS-388 in Combination with Toripalimab

SUMMARY:
This is a Phase 1/1b, open-label, first-in-human, dose-escalation and expansion study of CHS-388, a monoclonal antibody that targets IL-27, as a monotherapy and in combination in patients with solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/1b, open-label, first-in-human (FIH), dose-escalation and expansion study of CHS-388, a monoclonal antibody targeting IL-27, as a monotherapy and in combination in patients with solid tumors that will be conducted in 4 parts:

* Part A: CHS-388 monotherapy dose-escalation portion of the study will evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of CHS-388 as monotherapy in patients with advanced solid tumors.
* Part B: CHS-388 monotherapy expansion cohorts will evaluate the safety, efficacy, tolerability, PK, and pharmacodynamics of CHS-388 monotherapy in patients with advanced or metastatic ccRCC, advanced or metastatic HCC, and advanced or metastatic NSCLC in indication specific cohorts.
* Part C will evaluate the safety, preliminary efficacy, tolerability, and PK of CHS-388 in combination with pembrolizumab in patients with advanced RCC,HCC, or NSCLC.
* Part D will evaluate the safety, preliminary efficacy, tolerability, and PK of CHS-388 in combination with toripalimab in patients with advanced NSCLC.

ELIGIBILITY:
Part A and Part B Abbreviated Inclusion Criteria:

* ≥ 18 years of age
* Locally advanced or metastatic (Stage IV) solid tumor that has progressed during or after standard therapy, and for whom no available therapies are appropriate (based on investigator judgment)
* Patients in Part B with advanced or metastatic ccRCC, HCC, or NSCLC must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients with HCC in Part B must have at least 1 measurable target lesion according to modified RECIST (mRECIST)
* Patients with HCC must have unresectable disease, Barcelona Clinic Liver Cancer (BCLC1) Stage B (not eligible for transcatheter arterial chemoembolization [TACE]) or Stage C
* For patients in Part B with ccRCC, demonstrated progressive disease (PD) during or after the most recent treatment regimen. Prior treatment history must include progression during or after treatment with regimen(s) that have included a vascular endothelial growth factor (VEGF)-targeted agent and an immune checkpoint inhibitor. Patients who did not progress on but discontinued the VEGF-targeted agent for toxicity or intolerability are permitted.
* For patients in Part B with HCC, demonstrated PD during or after the most recent treatment regimen. Prior treatment history must include progression during or after treatment with a VEGF-targeted agent. Patients who did not progress on but discontinued the VEGF-targeted agent for toxicity or intolerability are permitted.
* For Part B patients in the tumor biopsy subsets only, must have tumor tissue that is accessible for pretreatment and on-treatment tumor biopsy in the opinion of the Investigator and be willing to undergo pretreatment and on-treatment biopsies per protocol
* Serum creatinine clearance ≥ 30 mL/min per Cockcroft-Gault formula or serum creatinine ≤ 2.0 x the upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN if elevated because of Gilbert's syndrome and ≤ 2 x ULN for patients with HCC or patients with known liver metastases)
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) < 2.5 x ULN (< 5 x ULN if liver metastasis or for patients with HCC)
* For patients with HCC, Child-Pugh class A or B7 with a serum albumin ≥ 2.8 g/dL (≥ 28 g/L)
* Adequate hematologic function, defined as absolute neutrophil count (ANC) ≥ 1.0 x 109/L, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100 x 109/L. For patients with HCC, platelet count ≥ 75 x 109/L without transfusion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients with NSCLC must have histologically confirmed locally advanced and/or metastatic Stage IV NSCLC
* Patients with NSCLC must have demonstrated progressive disease during or after the most recent treatment regimen

Part C Abbreviated Inclusion Criteria:

* ≥ 18 years of age
* Advanced RCC of any histology or advanced HCC previously treated with at least one systemic anticancer therapy OR histologically or cytologically confirmed metastatic or unresectable adenocarcinoma or squamous cell NSCLC
* Patients with HCC must have unresectable disease, Barcelona Clinic Liver Cancer (BCLC) Stage B (not eligible for transcatheter arterial chemoembolization) or Stage C
* At least 1 measurable lesion per RECIST 1.1
* Patients with HCC must have at least 1 measurable target lesion according to modified RECIST (mRECIST)
* ECOG performance status of 0-1
* ANC ≥1500/µL (1.5 x 109/L)
* Platelets ≥100 000/µL (≥ 100 x 109/L)
* Hemoglobin for participants with RCC: ≥9.0 g/dL; for participants with HCC: ≥8.5 g/dL
* Creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Total bilirubin ≤1.5 × ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* For patients with HCC, Child-Pugh Class A or B7 with a serum albumin ≥ 2.8 g/dL (≥ 28 g/L)
* Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study drug period (or beginning 14 days before the initiation of pembrolizumab for oral contraception), including 75 days after the last dose of CHS-388 or 120 days after the last dose of pembrolizumab; male patients must refrain from donating sperm during this period. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception with spermicide. Azoospermic male patients and WCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, female patients must still undergo pregnancy testing as described in this section.

Part C Abbreviated Inclusion Criteria Specific to Patients with RCC or HCC from Part A or Part B:

* Progressed on CHS-388 by RECIST 1.1
* Did not experience prior Grade ≥ 3 toxicity related to CHS-388
* Willingness to undergo pretreatment core or excisional biopsy if deemed safe and tumor is accessible, in the opinion of the Investigator
* Has received no systemic anticancer therapies between CHS-388 doses

Part C Abbreviated Inclusion Criteria specific to NSCLC Patients:

* No more than 3 prior lines of systemic therapy for unresectable or metastatic disease with prior radiologic progression on or following platinum-based chemotherapy and prior anti-PD-(L)1 therapy whether given alone or in combination

Part A and Part B Abbreviated Exclusion Criteria:

* Previously received an anti-IL-27 antibody or anti-IL-27 targeted therapy
* For patients in Part B with renal cell carcinoma (RCC), non-clear cell RCC histology
* For patients with HCC, known fibrolamellar or mixed hepatocellular cholangiocarcinoma
* History of Grade 4 allergic or anaphylactic reaction to any monoclonal antibody therapy or any excipient in the study drugs
* Major surgery within 4 weeks prior to Screening
* Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study

Part C Abbreviated Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug
* Previously received an anti-IL 27 antibody or anti-IL 27 targeted therapy (exception to patients who received CHS-388 in Part A or Part B)
* No prior systemic therapy for unresectable or metastatic disease
* Received > 4 prior systemic regimens for unresectable or metastatic disease (prior PD-(L)1 inhibitors are allowed if the patient did not discontinue therapy due to ≥ Grade 3 drug-related toxicity)
* For patients with HCC, fibrolamellar histology or mixed hepatocellular cholangiocarcinoma
* For patients with HCC, moderate or severe ascites
* For patients with HCC, inability to undergo disease evaluation with triphasic computed tomography or magnetic resonance imaging because of contrast allergy or other contraindication
* For patients with HCC, imaging findings consistent with ≥ 50% liver occupation by HCC tumors
* History of Grade 4 allergic or anaphylactic reaction to any monoclonal antibody therapy or any excipient in the study drugs
* Surgeries that required general anesthesia must be completed at least 2 weeks before first study drug administration
* Prior autologous stem cell transplant ≤ 3 months before the first dose
* Prior allogeneic hematopoietic cell transplant within 6 months of the first dose or with a history of or current clinical Graft-Versus-Host Disease
* Has had an allogenic tissue/solid organ transplant
* Other unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study

Part D Abbreviated Inclusion Criteria

* ≥ 18 years of age
* Histologically or cytologically confirmed metastatic or unresectable adenocarcinoma or squamous cell NSCLC
* No more than 3 prior lines of systemic therapy for unresectable or metastatic disease with prior radiologic progression on or following platinum-based chemotherapy and prior anti-PD-(L)1 therapy whether given alone or in combination
* At least 1 measurable lesion per RECIST 1.1
* ECOG performance status of 0-1
* ANC ≥1500/µL (1.5 x 109/L)
* Platelets ≥100 000/µL (≥ 100 x 109/L)
* Hemoglobin for participants with RCC: ≥9.0 g/dL
* Creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Total bilirubin ≤1.5 × ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study drug period (or beginning 14 days before the initiation of pembrolizumab for oral contraception), including 75 days after the last dose of CHS-388 or 180 days after the last dose of toripalimab; male patients must refrain from donating sperm during this period. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception with spermicide. Azoospermic male patients and WCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, female patients must still undergo pregnancy testing as described in this section.

Part D Abbreviated Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug
* Previously received an anti-IL 27 antibody or anti-IL 27 targeted therapy (exception to patients who received CHS-388 in Part A or Part B)
* No prior systemic therapy for unresectable or metastatic disease
* Received > 4 prior systemic regimens for unresectable or metastatic disease (prior PD-(L)1 inhibitors are allowed if the patient did not discontinue therapy due to ≥ Grade 3 drug-related toxicity)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a ≥ Grade 3 irAE.

because of contrast allergy or other contraindication

* History of Grade 4 allergic or anaphylactic reaction to any monoclonal antibody therapy or any excipient in the study drugs
* Surgeries that required general anesthesia must be completed at least 2 weeks before first study drug administration
* Prior autologous stem cell transplant ≤ 3 months before the first dose
* Prior allogeneic hematopoietic cell transplant within 6 months of the first dose or with a history of or current clinical Graft-Versus-Host Disease
* Has had an allogenic tissue/solid organ transplant
* Other unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
[Part A] Dose Limiting Toxicity (DLT) | Assessed during first 28 days of treatment
  Evaluation of DLT of CHS-388 as a monotherapy.
[Part B] Confirmed objective response rate (ORR) | Up to 24 months
  ORR will be estimated by the percentage of patients achieving a best overall response of CR or PR per RECIST v1.1 and iRECIST.
[Part C] DLT | Assessed during first 21 days of treatment
  Evaluation of DLT of CHS-388 in combination with pembrolizumab.
[Part C] Summary of adverse events (AEs) based on treatment emergent AEs (TEAEs) | Up to 24 months
  Safety and tolerability of CHS-388 + pembrolizumab will be assessed by summarizing AEs and will be based on TEAEs. A TEAE is an AE that emerges or worsens in the period from the first dose of study treatment to 30 days after the last dose of study drug assessed by per CTCAE version 5.0 or higher.
[Part C -NSCLC Cohort] Objective response rate (ORR) | Up to 24 months
  ORR will be estimated by the percentage of patients achieving a best overall response of CR or PR per RECIST v1.1 and iRECIST.
[Part D] Objective response rate (ORR) | Up to 24 months
  CR or PR per RECIST v1.1

SECONDARY OUTCOMES:
[Part A, Part B] Safety Analysis: Summary of adverse events (AEs) and based on treatment-emergent AEs (TEAEs) | Up to 24 months
  Safety and tolerability of CHS-388 will be assessed by summarizing adverse events (AEs) and will be based on treatment-emergent AEs (TEAEs).
[Part A, Part B, Part C] Pharmacokinetics (PK) of CHS-388 | Up to 24 months
  Serum concentrations of CHS-388 will be collected and analyzed to evaluate the PK of CHS-388.
[Part D] Pharmacokinetics (PK) of CHS-388 and toripalimab | Up to 24 months
  Serum concentrations of CHS-388 and toripalimab will be collected and analyzed to evaluate the PK of CHS-388 and toripalimab
[Part A, Part B] Pharmacodynamics of CHS-388 (pSTAT levels) | Up to 24 months
  Pharmacodynamics of CHS-388 will be evaluated in immune cell subsets via whole blood.
[Part A, Part C] Objective response rate (ORR) | Up to 24 months
  ORR will be estimated by the percentage of patients achieving a best overall response of CR or PR per RECIST v1.1 and iRECIST.
[Part A, Part B, Part C, Part D] Duration of response (DoR) | Up to 24 months
  DoR is defined as the time from the first documented response (CR or PR) to documented disease progression as determined by applicable disease criteria, or documented death due to any cause, whichever occurs first.
[Part A, Part B, Part C, Part D] Disease control rate (DCR) | Up to 24 months
  DCR is defined as the percentage of patients with CR, partial PR, or stable disease lasting a minimum of 12 weeks.
[Part A, Part B, Part C, Part D] Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from the first treatment on study with study drug to documented disease progression as determined by applicable disease criteria or death.
[Part C, Part D] Serum concentration of EBI3 | Up to 24 months
  Serum will be collected to assess EBI3 correlation with outcomes.
[Part C] Anti-drug Antibodies (ADAs) to CHS-388 | Up to 24 months
  Serum will be collected and assessed for the development of ADAs to CHS-388.
[Part D] Anti-drug Antibodies (ADAs) to CHS-388 and toripalimab | Up to 24 months
  Serum will be collected and assessed for the development of ADAs to CHS-388 and toripalimab.
[Part C - NSCLC Cohort] Summary of adverse events (AEs) based on treatment emergent AEs (TEAEs) | Up tp 24 months
  Safety and tolerability of CHS-388 + pembrolizumab will be assessed by summarizing AEs and will be based on TEAEs.
[Part D] Summary of adverse events (AEs) based on treatment emergent AEs (TEAEs) | Up tp 24 months
  Safety and tolerability of CHS-388 + toripalimab will be assessed by summarizing AEs and will be based on TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Koho Iizuka, MD, Study Chair — Coherus BioSciences
Locations (23):
- United States (18):
  - City of Hope, Duarte, California
  - University of Southern California (USC) - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Miami Leonard M. Miller School of Medicine (UMMSM), Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System (UMHS), Ann Arbor, Michigan
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Roswell Park, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC) - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center (University of Pittsburgh Cancer Institute (UPCI)), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Washington, Seattle, Washington
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore (NCCS), Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No